CLINICAL TRIAL: NCT07266168
Title: Efficacy and Safety of Ivarmacitinib in the Treatment of Patients With Polymyalgia Rheumatica: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: Efficacy and Safety of Ivarmacitinib in the Treatment of Patients With Polymyalgia Rheumatica
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: First Affiliated Hospital of Ningbo University (Network); Jinhua Central Hospital (Other); First People's Hospital of Hangzhou (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Huzhou Central Hospital (Other); Ningbo Medical Center Lihuili Hospital (Other Government); The Second Affiliated Hospital of Jiaxing University (Other); Affiliated Hospital of Jiaxing University (Other); Changxing People's Hospital (Other); Shanghai Zhongshan Hospital (Other); Ruijin Hospital (Other); Qilu Hospital of Shandong University (Other); The First Affiliated Hospital of Nanchang University (Other); RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-200
Record Dates: First submitted 2024-12-22; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Polymyalgia Rheumatics (PMR)
MeSH Terms: interventions — ivarmacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): The placebo group received a matched placebo for Ivarmacitinib treatment up to week 12. At week 12, the trial was unblinded, and the placebo group was switched to receive Ivarmacitinib treatment up to week 48, followed by a 4-week safety follow-up period up to week 52.
  Interventions: Drug: Ivarmacitinib tablet; Drug: placebo for lvarmacitinib
- Ivarmacitinib tablet (Active Comparator): The treated group received Ivarmacitinib at 4 mg/day for 48 weeks, followed by a 4-week safety follow-up period up to week 52.
  Interventions: Drug: Ivarmacitinib tablet

INTERVENTIONS:
Drug: Ivarmacitinib tablet — Targets JAK kinases to block signal transduction of the JAK-STAT pathway
Drug: placebo for lvarmacitinib — Treatment using blank placebo
  Arms: placebo

SUMMARY:
The study intends to explore the efficacy and safety of Ivarmacitinib in therapy for polymyalgia rheumatica through a multicenter, randomized, double-blind, placebo-controlled study, and to explore the effectiveness of Ivarmacitinib as an oral glucocorticoid-sparing alternative in the treatment of polymyalgia rheumatica.

DETAILED DESCRIPTION:
This study plans to enroll 80 patients with clinically confirmed severe active polymyalgia rheumatica. After enrollment, participants will be randomly assigned in a 1:1 ratio to either the experimental group or the placebo group. All patients will receive a single dose of long-acting glucocorticoid in Week 1. Both groups will continue their assigned treatment until Week 12, when unblinding will occur. Thereafter, the placebo group will switch to ivarmacitinib, and both groups will continue treatment until Week 48, followed by a 4-week safety follow-up period until Week 52.

ELIGIBILITY:
Inclusion Criteria:

1. Age and Weight: 50-75 years old, body weight 40-80 kg.
2. Diagnosis: Confirmed diagnosis of polymyalgia rheumatica (PMR) according to the 2012 ACR/EULAR classification criteria .
3. Disease Activity: CRP-PMR-AS (C-reactive protein polymyalgia rheumatica activity score) ≥17 .
4. Glucocorticoid Use:

   * Newly Diagnosed Patients: No glucocorticoid use within 12 weeks prior to enrollment.
   * Relapsed Patients: No increase in glucocorticoid dosage within 2 weeks prior to enrollment, and willingness to discontinue current glucocorticoids after enrollment.
5. Compliance: Participants must understand and agree to adhere to study procedures and restrictions.

   -

Exclusion Criteria:

1. Allergy: Known hypersensitivity to the investigational drug or excipients (including lactose, cellulose-lactose, low-substituted hydroxypropyl cellulose (L-HPC), colloidal silicon dioxide, stearic acid).
2. Comorbidities:

   * Giant cell arteritis (GCA) .
   * Other diffuse connective tissue diseases (e.g., systemic lupus erythematosus), spondyloarthropathy, or active fibromyalgia .
3. Uncontrolled Chronic Conditions:

   * Diabetes (HbA1c ≥8.0%) or uncontrolled hypertension (resting SBP ≥140 mmHg and/or DBP ≥90 mmHg) .
   * Clinically significant ECG abnormalities (e.g., acute myocardial ischemia, myocardial infarction, severe arrhythmia, QTc >500 ms).
4. Organ Dysfunction:

   * Liver/Kidney Impairment:
   * AST/ALT ≥2× upper limit of normal (ULN).
   * Serum creatinine or total bilirubin ≥1.5× ULN .
5. Malignancy: History of malignancy within the past 5 years.
6. Infections:

   * Active uncontrolled infections (e.g., tuberculosis, hepatitis B surface antigen (HBsAg) positive with elevated HBV-DNA, HCV, HIV, or active syphilis).
   * Severe herpes zoster infection or systemic antimicrobial therapy within 2 weeks prior to randomization.
7. Reproductive Plans: Pregnancy planning within 1 year.
8. Prior Medications: Previous use of JAK inhibitors.
9. Thrombosis: History of thrombotic events.
10. Other: Any condition deemed inappropriate by the investigator for participation in this clinical study.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with CRP PMR-AS ≤10 at Week 12 without oral glucocorticoid use from Week 0 to Week 12; | up to 12 weeks
  The proportion of patients with CRP PMR-AS ≤10 at Week 12 without oral glucocorticoid use from Week 0 to Week 12

SECONDARY OUTCOMES:
Proportion of Patients Achieving CRP-PMR-AS ≤10 Without Oral Glucocorticoids | up to 48 weeks
  Measured at Weeks 16, 20, 28, 36, and 48.
Erythrocyte sedimentation rate (ESR) | up to 48 weeks
  Changes in Inflammatory Markers
level of C-reactive protein (CRP) | up to 48 weeks
  Markers: C-reactive protein (CRP).
level of Interleukin-6 (IL-6). | up to 48 weeks
  Cytokine: Interleukin-6 (IL-6).
Cumulative Glucocorticoid Dose at Week 48. | up to 48 weeks
  Long-Term Follow-Up Outcome
Relapse Rate at Week 48 in Both Groups | up to 48 weeks
  Relapse Definition: PMR-AS ≥10 AND requiring escalation of glucocorticoid therapy based on the original regimen.